CLINICAL TRIAL: NCT05264857
Title: Decision Aid for Management of Thyroid Nodules and Early Thyroid Cancer
Brief Title: Decision Aid and Thyroid Nodules Management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Lukasz Czerwonka, Head and Neck Surgeon, Stony Brook University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SBU-DECISION-AID-THYROID
Record Dates: First submitted 2022-02-17; First posted 2022-03-03 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Thyroid Nodule
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Thyroid nodule information (Experimental)
  Interventions: Behavioral: Thyroid Nodule Management Education

INTERVENTIONS:
Behavioral: Thyroid Nodule Management Education — Participants will receive information about thyroid nodules and their management

SUMMARY:
Patients with small favorable malignant or indeterminate thyroid nodules will receive information about management of thyroid nodules. Participants will be asked to complete brief surveys at the time of enrollment, shortly after the consultation appointment with the surgeon, and a few months after either the consultation or the surgery, to assess their satisfaction with their decision and decision making process. All participants will receive routine care and counseling by their endocrinologist and surgeon.

ELIGIBILITY:
Inclusion Criteria:

* Histology showing indeterminate or malignant thyroid pathology (Bethesda III-VI)
* Thyroid nodule size less or equal to 2cm

Exclusion Criteria:

* History of thyroid surgery
* History of thyroid cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2022-02-08 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Rate of congruence between informed values and treatment choice | 6 months from surgery or surgical consultation date
  Percent of patients with congruence between treatment option and informed values based on a survey

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Czerwonka, MD, Principal Investigator — Lukasz.Czerwonka@stonybrookmedicine.edu
Locations (1):
- Stony Brook University Cancer Center, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No